CLINICAL TRIAL: NCT01112436
Title: The Effect of Periarticular Injection of Multi-drug Regimen on Pain in Patient Receiving Partial Hip Replacement:Randomized Prospective Study.
Brief Title: The Effect of Periarticular Multi-Drug Regimen on Pain After Partial Hip Replacement
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other)
Responsible Party: Yong Chan Ha, Chung-Ang University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ChunaAngUH
Record Dates: First submitted 2010-04-22; First posted 2010-04-28 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2010-04

CONDITIONS: Femoral Neck Fracture
Keywords: Pain; preemptive; Postoperative; delirium
MeSH Terms: conditions — Femoral Neck Fractures; Pain; Delirium

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- control group (group C) (Placebo Comparator): control group will receive no medication preoperatively and during operation
  Interventions: Drug: none of medication preoperatively and intraoperatively
- periarticular injecion group (group I) (Active Comparator): patients in Group I will receive oral oxycodone SR 10 mg and celecoxib 200 mg 1 hour preoperatively with sips of water, and receive periarticular injection of combination of ropivacaine 15 mg, morphine 10 mg, ketorolac 30 mg epinephrine 0.3 mg and cefmetazole 1000mg during operation.
  Interventions: Drug: periarticular injection of multidrug regimen

INTERVENTIONS:
Drug: periarticular injection of multidrug regimen — periarticular injection of combination of ropivacaine 15 mg, epinephrine 0.3mg, cefmetazole 1000mg, ketorolac 30mg, morphine HCL 10 mg
  Other Names: injection near the hip joint
  Arms: periarticular injecion group (group I)
Drug: none of medication preoperatively and intraoperatively — Patients in Group C wil receive none of medication preoperatively and intraoperatively
  Other Names: Patients in Group C wil receive none of medication
  Arms: control group (group C)

SUMMARY:
This prospective randomized study aims to evaluate the effectiveness of periarticular multi-drug regimen injection on the relief of pain in patients undergoing partial hip replacement.

Total 258 patients will be randomized into one of two groups (groupC or groupI) based on Excel number generation.

Patients in group C will receive no medication intraoperatively, and patients in group I will receive oral oxycodone and celecoxib preoperatively and a periarticular injection of multi-drug regimen during operation.

Visual analogue scale pain scores, fentanyl consumption and the frequency at which patients pushed the button (FPB) of a patient-controlled analgesia system will be recorded at 1, 4, 7 postoperative day.

DETAILED DESCRIPTION:
Patients in group I will receive oxycodone SR 10 mg, and celecoxib 200 mg with 10 ml of water 1 hour before surgery.

And patients in group I will receive periarticular injection of 50 ml solution which contains ropivacaine 15 mg, epinephrine 0.3 mg, cefmetazole 1000mg, ketorolac 30 mg and morphine HCL 10mg before closure of surgical wound.

Patients in group C will receive no medication.

ELIGIBILITY:
Inclusion Criteria:

* femoral neck fracture
* partial hip replacement

Exclusion Criteria:

* r/o infection
* reoperation
* mental change

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 258 (Estimated)
Dates: Start 2010-05; Primary Completion 2012-04 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale 1day | Post Op 1 day
  Patients will be assessed for pain using a visual analogue pain scale (VAS). It is usually a horizontal line, 100 mm in length, anchored by word descriptors at each end; left side end which represents 0 is 'No pain', right side end with 100 is 'Very severe pain'. The patient marks on the line the point that they feel represents their perception of their current state. The VAS score is determined by measuring in millimeters from the left hand end of the line to the point that the patient marks.
  To check the severity of pain VAS will be measured at post op 1day.

SECONDARY OUTCOMES:
Opioid consumption 1day | Post Op 1 day
  The patients will be taught to push the button of the PCA system, which delivered a bolus of drug, each time pain occurred. In the case of persistent pain greater than a visual analogue scale (VAS) pain score of 30 mm, an additional 50 μg of fentanyl will be injected intra-venously by nursing staff until the pain was relieved to a level less than a VAS pain score of 30 mm. And sum of delivery from PCA system and additional opioid fom immediately after operation to post op 1daywill be measured.
FPB 1day | Post Op 1 day
  The patients will be taught to push the button of the PCA system, which delivered a bolus of drug, each time pain occurred. And total frequency of patient to push the button of the PCA machine (FPB) fom immediately after operation to post op 1day will be measured.
delirium rating scale at admission | at admission
  Delirium rating scale wiil be measured to compare with the post op delerium scale at admisssion.
Visual Analogue Scale 4day | Post OP 4day
  Patients will be assessed for pain using a visual analogue pain scale (VAS). It is usually a horizontal line, 100 mm in length, anchored by word descriptors at each end; left side end which represents 0 is 'No pain', right side end with 100 is 'Very severe pain'. The patient marks on the line the point that they feel represents their perception of their current state. The VAS score is determined by measuring in millimeters from the left hand end of the line to the point that the patient marks.
  To check the severity of pain VAS will be measured at post op 4day.
Visual Analogue Scale 7day | Post Op 7day
  Patients will be assessed for pain using a visual analogue pain scale (VAS). It is usually a horizontal line, 100 mm in length, anchored by word descriptors at each end; left side end which represents 0 is 'No pain', right side end with 100 is 'Very severe pain'. The patient marks on the line the point that they feel represents their perception of their current state. The VAS score is determined by measuring in millimeters from the left hand end of the line to the point that the patient marks.
  To check the severity of pain VAS will be measured at post op 7day.
Opioid consumption 4day | Post Op 4 day
  The patients will be taught to push the button of the PCA system, which delivered a bolus of drug, each time pain occurred. In the case of persistent pain greater than a visual analogue scale (VAS) pain score of 30 mm, an additional 50 μg of fentanyl will be injected intra-venously by nursing staff until the pain was relieved to a level less than a VAS pain score of 30 mm. And sum of delivery from PCA system and additional opioid fom post op 1day to post op 4 day will be measured.
Opioid consumption 7day | Post Op 7 day
  The patients will be taught to push the button of the PCA system, which delivered a bolus of drug, each time pain occurred. In the case of persistent pain greater than a visual analogue scale (VAS) pain score of 30 mm, an additional 50 μg of fentanyl will be injected intra-venously by nursing staff until the pain was relieved to a level less than a VAS pain score of 30 mm. And sum of delivery from PCA system and additional opioid fom post op 4day to post op 7 day will be measured.
FPB 4day | Post Op 4 day
  The patients will be taught to push the button of the PCA system, which delivered a bolus of drug, each time pain occurred. And total frequency of patient to push the button of the PCA machine (FPB) fom post op 1day to post op 4 day will be measured.
FPB 7day | Post Op 7 day
  The patients will be taught to push the button of the PCA system, which delivered a bolus of drug, each time pain occurred. And frequency of patient to push the button of the PCA machine (FPB) fom post op 4day to post op 7day will be measured.
delirium rating scale 1day | Post Op 1day
  Delirium rating scale wiil be measured to check the incidence and severity of delirium at post-op 1day.
delirium rating scale 4day | Post Op 4day
  Delirium rating scale wiil be measured to check the incidence and severity of delirium at post-op 4day.
delirium rating scale 7day | Post Op 7day
  Delirium rating scale wiil be measured to check the incidence and severity of delirium at post-op 7day.

CONTACTS AND LOCATIONS:
Overall Officials: Yong Chan Ha, M.D. & Ph.D., Study Director — Chung-Ang University Hosptial, Chung-Ang University College of Medicine; Hyun Kang, M.D. & Ph.D., Principal Investigator — Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Locations (1):
- ChungAng University, Seoul, South Korea